CLINICAL TRIAL: NCT06603493
Title: The Silent Saboteur: The Impact of Headaches on Sleep Disorders, Central Sensitization, Depression, Anxiety and Stress
Brief Title: Headaches: Effects on Sleep, Sensitization, and Psychological Factors
Status: Completed | Type: Observational
Sponsor: Nagihan Acet (Other)
Responsible Party: Sponsor-Investigator, Nagihan Acet, Asst. Prof., Atılım University
Organization: Atılım University (Other)
Other Study IDs: Atılım Physiotherapy
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Headache Disorder
Keywords: Headache; sleep; Central Nervous System Sensitization; Depression; Anxiety; Pain
MeSH Terms: conditions — Headache Disorders; Headache; Depression; Anxiety Disorders; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Headache Group: individuals diagnosed with migraine and tension-type headache according to the International Classification of Headache Disorders (International Classification of Headache Disorders, 3rd edition) will be placed in the headache group
  Interventions: Other: Assessment of sleep disorders; Other: Assessment of Central Sensitization; Other: Assessment of depression, anxiety and stress levels
- Control Group: Individuals aged 18-65 without headaches will be placed in control group.
  Interventions: Other: Assessment of sleep disorders; Other: Assessment of Central Sensitization; Other: Assessment of depression, anxiety and stress levels

INTERVENTIONS:
Other: Assessment of sleep disorders — : Sleep disturbances will be assessed with the Pittsburgh Sleep Quality Index
Other: Assessment of Central Sensitization — Central sensitization will be assessed with the Central Sensitization Inventory
Other: Assessment of depression, anxiety and stress levels — Depression, anxiety and stress levels will be assessed using the Depression, Anxiety, Stress Scale (DASS-21)

SUMMARY:
Headache is one of the most common health problems in the society and negatively affects the quality of life of individuals. Increasing complaints of headache in recent years can be associated with many physiological and psychological factors. Sleep disturbances are one of these factors. Inadequate or non-restful sleep can interfere with the normal course of physical, mental, social and emotional functions. Impaired sleep quality interferes with the body's process of repairing and regenerating itself, which can lead to more serious health problems in the long term. Secondly, headaches can also lead to neurophysiological changes such as central sensitization. Central sensitization causes the nervous system to become hypersensitive, lowering the pain threshold and increasing pain perception. Finally, headache can have psychological effects by increasing levels of depression, anxiety and stress.

This study aimed to determine the effects of headache on sleep disturbances, central sensitization, depression, anxiety and stress.

DETAILED DESCRIPTION:
Headache is one of the most common health problems in the society and types of headache have a significant negative impact on the quality of life of individuals. Headaches can occur in a wide range from temporary discomfort to chronic problems and can negatively affect individuals' work performance, social life and general health . In recent years, complaints of headache have been increasing in the society. This may be associated with factors such as stress factors of modern life, sleep irregularities and increased use of technology.

One of the factors most affected by headache is sleep disturbance. Especially the presence of migraine can lead to sleep disorders. Sleep disorders consist of various conditions that disrupt normal sleep patterns and are one of the most common problems encountered in clinical practice. Inadequate or non-restful sleep may interfere with the normal course of physical, mental, social and emotional functions. Impaired sleep quality inhibits the body's process of self-repair and regeneration, which can lead to more serious health problems in the long term.

Establishing the relationship between sleep and headache can make a significant contribution to the management of headache.

Headaches can also be an important trigger of central sensitization. Central sensitization is an adaptive, activity-dependent and dynamic neurophysiological phenomenon]. This process involves neurobiological changes in neurons in the dorsal horn of the spinal cord.]. These changes include increased excitability, enhanced synaptic transmission and decreased inhibition. In summary, central sensitization is a condition in which the nervous system becomes hypersensitive and pain is perceived as more severe than normal. Especially in individuals with chronic headache, central sensitization may develop as a result of continuous stimulation of the nervous system and this may lead to a decrease in pain threshold and an increase in pain perception. Especially the fact that chronic headache triggers central sensitization is a factor that makes the treatment process very difficult and this situation seriously affects the quality of life of patients.

The psychological effects of headache cannot be ignored. Headache can increase depression, anxiety and stress levels. When pain becomes a constant source of anxiety, it makes it difficult to perform daily activities and negatively affects the general mood of the person. Depression and anxiety can increase the severity of headaches, and headaches can trigger these psychological conditions. Stress can be both a cause and a consequence of headache; especially tension-type headaches are closely related to stress. Therefore, it is important to consider the psychological status in the treatment of headache.

The presence of headache may affect many factors such as sleep disturbance, central sensitization, depression, anxiety and stress, and revealing these effects will contribute to the development of treatment approaches in headache treatment.

In the light of the above information, the aim of the present study was to determine the effect of the presence of headache on sleep disorders, central sensitization, depression, anxiety and stress.

ELIGIBILITY:
Inclusion Criteria:

* being 18-65 years who agreed to participate

Exclusion Criteria:

* Neurological disorders
* Musculoskeletal diseases
* Chronic pain conditions
* Psychiatric diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-65 with and without headaches.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Assessment of sleep disorders | baseline
  : Sleep disturbances were assessed with the Pittsburgh Sleep Quality Index (PSQI) . The PSQI is a 19-question questionnaire used to measure sleep habits over the past month and has 7 components. The total score ranges from 0 to 21, with higher scores indicating poor sleep quality. Scores of 5 and above are considered as sleep disturbance.
Assessment of depression, anxiety and stress levels | baseline
  Depression, anxiety and stress levels were assessed using the Depression, Anxiety, Stress Scale (DASS-21). The DASS-21 consists of depression, anxiety and stress subscales, each with 7 questions. A maximum of 42 points can be obtained for each component (the first score is multiplied by two). Higher scores indicate the severity of the respective disorder. Cut-off values are different for each disorder: for depression, 0-9 (normal) to 28 and above (very severe), for anxiety 0-7 (normal) to 20 and above (very severe), and for stress 0-14 (normal) to 34 and above (very severe).
Assessment of Central Sensitization | baseline
  Central sensitization was assessed with the Central Sensitization Inventory (SSI.) The SSE consists of 25 questions. The total score ranges from 0 to 100 and a score of 40 and above indicates the presence of central sensitization.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sariçam, H., The psychometric properties of Turkish version of Depression Anxiety Stress Scale-21 (DASS-21) in health control and clinical samples. Journal of Cognitive Behavioral Psychotherapies and Research, 2018. 7(1): p. 19.
- [Result] Lovibond, S.H., Manual for the depression anxiety stress scales. Sydney psychology foundation, 1995.
- [Result] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Result] Duzce Keles E, Birtane M, Ekuklu G, Kilincer C, Caliyurt O, Tastekin N, Is EE, Ketenci A, Neblett R. Validity and reliability of the Turkish version of the central sensitization inventory. Arch Rheumatol. 2021 Oct 18;36(4):518-526. doi: 10.46497/ArchRheumatol.2022.8665. eCollection 2021 Dec. PMID 35382371
- [Result] Ağargün, M.Y., H. Kara, and Ö. Anlar, The validity and reliability of the Pittsburgh Sleep Quality Index. Turk Psikiyatri Derg, 1996. 7(2): p. 107-15.
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Pambudi, P. and O. Sidabutar, Correlation between the Degree of Psychological Stress with Pain Intensity in Tension-Type Headache Patients. Jurnal Kedokteran Brawijaya, 2024: p. 6-10.
- [Result] Suzuki K, Suzuki S, Shiina T, Kobayashi S, Hirata K. Central Sensitization in Migraine: A Narrative Review. J Pain Res. 2022 Sep 7;15:2673-2682. doi: 10.2147/JPR.S329280. eCollection 2022. PMID 36101891
- [Result] Sebastianelli G, Casillo F, Abagnale C, Renzo AD, Cioffi E, Parisi V, Lorenzo CD, Fazio F, Petricola F, Mattia C, Serrao M, Schoenen J, Coppola G. Central sensitization mechanisms in chronic migraine with medication overuse headache: a study of thalamocortical activation and lateral cortical inhibition. Cephalalgia. 2023 Oct;43(10):3331024231202240. doi: 10.1177/03331024231202240. PMID 37795647
- [Result] van Griensven H, Schmid A, Trendafilova T, Low M. Central Sensitization in Musculoskeletal Pain: Lost in Translation? J Orthop Sports Phys Ther. 2020 Nov;50(11):592-596. doi: 10.2519/jospt.2020.0610. PMID 33131390
- [Result] Karna B, Sankari A, Tatikonda G. Sleep Disorder. 2023 Jun 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560720/ PMID 32809555
- [Result] Stovner LJ, Hagen K, Linde M, Steiner TJ. The global prevalence of headache: an update, with analysis of the influences of methodological factors on prevalence estimates. J Headache Pain. 2022 Apr 12;23(1):34. doi: 10.1186/s10194-022-01402-2. PMID 35410119
- [Result] R P, S C N, S H, K R. Migraine Disability, Quality of Life, and Its Predictors. Ann Neurosci. 2020 Jan;27(1):18-23. doi: 10.1177/0972753120929563. Epub 2020 Jul 3. PMID 32982095
- [Result] Abu Bakar N, Tanprawate S, Lambru G, Torkamani M, Jahanshahi M, Matharu M. Quality of life in primary headache disorders: A review. Cephalalgia. 2016 Jan;36(1):67-91. doi: 10.1177/0333102415580099. Epub 2015 Apr 17. PMID 25888584
- [Result] Stovner LJ, Andree C. Prevalence of headache in Europe: a review for the Eurolight project. J Headache Pain. 2010 Aug;11(4):289-99. doi: 10.1007/s10194-010-0217-0. Epub 2010 May 16. PMID 20473702